CLINICAL TRIAL: NCT06423417
Title: LifeHack: RCT Evaluating the Effectiveness of a Guided E-health Programme in Improving Mental Wellbeing in University Students.
Brief Title: RCT: the Effectiveness of LifeHack in Improving Mental Wellbeing in University Students.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Collaborators: Maastricht University (Other); VU University of Amsterdam (Other); Utrecht University (Other); University of Amsterdam (Other); Rotterdam University of Applied Sciences (Other); Erasmus University Rotterdam (Other); Avans University of applied sciences (Unknown); InHolland University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Sanne van Luenen, assistant professor in the Clinical Psychology unit at the Institute of Psychology, Universiteit Leiden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-10-30-S.vanLuenen-V1-506
Record Dates: First submitted 2024-05-08; First posted 2024-05-21 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-05

CONDITIONS: Internet-based Intervention; Waiting List Control Group; Depression; Anxiety; Stress; Quality of Life; Mental Wellbeing; Resilience
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The present study is a two-arm randomized controlled superiority trial. This trial will be conducted in a university setting. A guided web-based resilience and mental wellbeing programme (LifeHack) will be compared to a waiting list condition. Participants in the waiting list condition will start with the programme 4 weeks after randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LifeHack (Experimental): LifeHack is a guided (weekly feedback by a coach is provided) e-heath self-help application, which is based on cognitive behavioral techniques. The goal of LifeHack is to improve mental wellbeing.
  The guided internet-based self-help programme LifeHack was developed based on existing literature and adapted in collaboration with university students. The programme comprises twelve modules that are delivered via computer, laptop, tablet, or mobile phone. The modules take approximately 30 minutes on 4 themes (mood management, productivity, self-worth and relationships).
  Guidance:
  E-coaches will be trained clinical psychology master students. E-coaches will provide asynchronous written personalized feedback to each participant through the program platform within 48 hours (counting workdays only) after session completion. The aim of the written feedback is to increase motivation and adherence of the participants.
  Interventions: Behavioral: LifeHack
- Control group (No Intervention): Participants in the waiting list control condition will start with the programme 4 weeks after randomization.

INTERVENTIONS:
Behavioral: LifeHack — See arm description
  Arms: LifeHack

SUMMARY:
Psychological issues are common among university students and affect mental wellbeing. The Caring Universities (CU) project, involving nine Dutch universities, aims to enhance students' mental health through an annual online questionnaire and a platform offering guided eHealth interventions. One intervention, LifeHack, utilizes cognitive behavioral therapy-based modules to improve mental wellbeing by enhancing resilience and life skills. The effects of LifeHack with pre-post measurements (total n = 216 at post-test) found found that LifeHack led to improvements in mental wellbeing, but dropout rates were influenced by lack of motivation and module relevance. A personalized version of LifeHack is being developed to address these issues and will be evaluated in an RCT to assess its effectiveness in improving mental wellbeing and related outcomes among university students.

DETAILED DESCRIPTION:
Psychological problems are prevalent among university students and are associated with lower mental wellbeing and resilience. Universities provide an excellent environment for students to enhance mental wellbeing, resilience, and acquire life skills.

Caring Universities (CU) is an internationally embedded consortium of nine Dutch universities aimed at improving students' mental wellbeing. The CU project consists of two components: 1) an annual online questionnaire assessing students' mental health; and 2) a platform offering free, guided eHealth interventions to enhance mental well-being.

One of the interventions on the CU platform - called LifeHack - seeks to enhance mental wellbeing by increasing resilience, teaching life skills, and strengthening mental wellbeing. LifeHack is a guided eHealth intervention based on cognitive behavioural therapy, comprising 13 modules of approximately 30 minutes each focusing on four themes (mood management, productivity, self-worth, and relationships). We investigated the effects of LifeHack with pre-post measurements (total n = 216 at post-test) and found that after following LifeHack, mental wellbeing improved with small to moderate effect sizes. Additionally, students reported satisfaction with the programme and the eCoach. However, participants indicated lack of motivation and early symptom reduction as important reasons for drop-out. Furthermore, the diverse topics covered in LifeHack may not be relevant to all students, leading to more dropouts.

Currently, there are two versions of LifeHack: one 'structured', where modules must be completed in order, and one 'free choice', where all modules are available from the start and none are mandatory. For the proposed study, the free choice version of LifeHack will be used and adapted in co-creation with students as follows: participants will be asked which topics they find most important and want to work on. Based on their answers, a personalized selection of modules will be presented, and students can choose which module to start with. Each module is standalone, allowing students to proceed to another module or stop after completing one or more. Each module has a clear structure, beginning with goal formulation and concluding with an action plan. The new adapted version of LifeHack will be personalized and tailored for each student, aiming to improve motivation and reduce dropout rates.

With the current study, we aim to examine the effectiveness of the adapted version of LifeHack in an RCT to enhance mental wellbeing in university students. Secondary objectives include investigating differences between the intervention and control groups on students' self-report questionnaire resilience scores, depression scores, anxiety scores, stress-related scores, and mental health quality of life scores (pretest vs post-test). Additional outcomes include satisfaction with the programme and the eCoach, as well as adherence to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being fluent in Dutch and/or English
* Being enrolled as a student at one of the 9 participating universities
* Being 16 years of age or older
* Having access to a PC or mobile device with internet access
* Provide informed consent before participation
* Score of 50 or lower on the MHC-SF. This is 1 SD above the mean baseline score of participants of LifeHack. This inclusion criterion ensures no students with optimal mental wellbeing are included because they will not be able to show any change.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Mental wellbeing (MHC-SF) | T0 (baseline), T1 (4 weeks post-baseline active group), T2 (4 weeks post-baseline wait list group), T3 (4 weeks post-T2 wait list group), T4 (6 months post-baseline both groups)
  Mental Health Continuum-Short Form, MHC-SF (Lamers et al., 2011).

SECONDARY OUTCOMES:
Resilience (BRS) | T0 (baseline), T1 (4 weeks post-baseline active group), T2 (4 weeks post-baseline wait list group), T3 (4 weeks post-T2 wait list group), T4 (6 months post-baseline both groups)
  Brief Resilience Scale (Smith et al., 2008).
Depressive symptoms (PHQ-9) | T0 (baseline), T1 (4 weeks post-baseline active group), T2 (4 weeks post-baseline wait list group), T3 (4 weeks post-T2 wait list group), T4 (6 months post-baseline both groups)
  Patient Health Questionnaire - 9, PHQ-9 (Kroenke et al., 2001).
Stress related symptoms (PSS-10) | T0 (baseline), T1 (4 weeks post-baseline active group), T2 (4 weeks post-baseline wait list group), T3 (4 weeks post-T2 wait list group), T4 (6 months post-baseline both groups)
  Perceived Stress Scale-10, PSS-10 (Cohen, 1988).
Symptoms of anxiety (GAD-7) | T0 (baseline), T1 (4 weeks post-baseline active group), T2 (4 weeks post-baseline wait list group), T3 (4 weeks post-T2 wait list group), T4 (6 months post-baseline both groups)
  Generalized Anxiety Disorder-7 scale, GAD-7 (Spitzer et al., 2006).
Quality of life (MHQoL) | T0 (baseline), T1 (4 weeks post-baseline active group), T2 (4 weeks post-baseline wait list group), T3 (4 weeks post-T2 wait list group), T4 (6 months post-baseline both groups)
  Mental Health Quality of Life questionnaire, MHQoL (Krugten et al., 2022).
Demographics | T0 (baseline)
  E.g. gender, age, nationality

OTHER OUTCOMES:
Depression and anxiety (PHQ-4) after each module. | After each module (approximately once per week)
  Patient Health Questionnaire - 4 (Kroenke et al., 2009). After each module, the PHQ-4 will be assessed in both groups.
Client satisfaction (CSQ-8) | 4 weeks post-baseline active group and 4 weeks post-T2 wait list group.
  The Client Satisfaction Questionnaire, CSQ-8 (Larsen et al., 1979)
E-coach evaluation (WAI-I) | 4 weeks post-baseline active group and 4 weeks post-T2 wait list group.
  We will also ask participants to evaluate the e-coach at the post-test. The questions about e-coach evaluation will be based on the Working Alliance Inventory for Guided Internet Interventions (WAI-I) (Gómez Penedo et al., 2020)
Adherence (Log info) | T1 (4 weeks post-baseline active group), T2 (4 weeks post-baseline wait list group), T3 (4 weeks post-T2 wait list group), T4 (6 months post-baseline both groups)
  Adherence will be measured by the total number of completed sessions, time spent on the platform, and the number of logins.

CONTACTS AND LOCATIONS:
Overall Officials: Sanne van Luenen, PhD, Principal Investigator — Leiden University
Locations (2):
- Netherlands (2):
  - VU Amsterdam, Amsterdam
  - Leiden University, Leiden

IPD SHARING:
Plan to Share IPD: No